CLINICAL TRIAL: NCT06821451
Title: A Prospective, Single-center, Non-inferiority Clinical Trial Study Evaluating the Effectiveness and Safety of Bronchoscopic Navigation Robot (bronchial Navigation Positioning Device) Guided Dye Marking-assisted Thoracoscopic Pulmonary Nodule Resection
Brief Title: Bronchoscopic Navigation Robot-guided Dye Marking-assisted Thoracoscopic Pulmonary Nodule Resection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hecheng Li M.D., Ph.D, Chair of Department of Thoracic Surgery, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTS-025
Record Dates: First submitted 2025-02-04; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Lung Nodules

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Active Comparator): Preoperative CT data creates a 3D image of the lung anatomy to plan the navigation path. The surgeon controls the robotic arm in real-time to reach staining marker points for pulmonary nodule localization. After placing the staining catheter in the working channel, 1 ml of indocyanine green is injected at the site. Then the patient is positioned laterally for video-assisted thoracoscopic surgery for nodule resection, initially focusing on sub-lobar resection. More extensive resection is determined based on intraoperative frozen section results.
  Interventions: Device: Bronchoscopic navigation robot
- Control group (Sham Comparator): Based on preoperative CT data, a three-dimensional image of the virtual bronchi is created to plan the navigation path, and manual registration is completed by selecting registration points using a conventional bronchoscope. After registration, the target position is reached under the guidance of the magnetic navigation positioning system, and when the positioning sensor indicates that it has arrived at the staining marker point, a staining catheter is inserted through the working channel to inject 1 ml of indocyanine green at the marker site, followed by thoracoscopic resection of the pulmonary nodule.
  Interventions: Device: Conventional electromagnetic navigation bronchoscope

INTERVENTIONS:
Device: Bronchoscopic navigation robot — Preoperative CT data creates a 3D image of the lung anatomy to plan the navigation path. The surgeon controls the robotic arm in real-time to reach staining marker points for pulmonary nodule localization. After placing the staining catheter in the working channel, 1 ml of indocyanine green is injected at the site. Then the patient is positioned laterally for video-assisted thoracoscopic surgery for nodule resection, initially focusing on sub-lobar resection. More extensive resection is determined based on intraoperative frozen section results.
  Other Names: bronchoscopic navigation positioning device; Robotic-assisted bronchoscopy; robotic-assisted bronchoscopy system
  Arms: Treatment group
Device: Conventional electromagnetic navigation bronchoscope — Based on preoperative CT data, a three-dimensional image of the virtual bronchi is created to plan the navigation path, and manual registration is completed by selecting registration points using a conventional electromagnetic bronchoscope. After registration, the target position is reached under the guidance of the magnetic navigation positioning system, and when the positioning sensor indicates that it has arrived at the staining marker point, a staining catheter is inserted through the working channel to inject 1 ml of indocyanine green at the marker site, followed by thoracoscopic resection of the pulmonary nodule.
  Other Names: ENB; Electromagnetic navigation bronchoscopy system
  Arms: Control group

SUMMARY:
With the widespread use of low-dose spiral CT screening for the lungs, an increasing number of small nodules are being detected, and surgical resection is the preferred method for clinical intervention of pulmonary nodules. Staining localization can assist surgeons in accurately locating pulmonary nodules during surgery, achieving complete resection of the nodules while minimizing the resection area, thereby optimizing surgical outcomes.

The study will include individuals with pulmonary nodules detected by CT scans who require color localization assistance for thoracoscopic pulmonary nodule resection, randomly divided into two groups: one group will receive bronchoscopic navigation-assisted staining localization, while the other group will receive staining localization guided by an electromagnetic navigation system. The primary outcome is to evaluate the success rate of staining localization between the two groups.

This study aims to assess, through a prospective, single-center, randomized controlled clinical trial, whether the success rate of staining localization guided by bronchoscopic navigation robots (experimental group) is not lower than that of staining localization guided by the electromagnetic navigation system (control group), while potentially offering advantages such as a shorter learning curve, ease of operation, and reduced surgical time. This will provide a new efficient and safe method for the localization of pulmonary nodules clinically, greatly supporting accurate treatment of pulmonary nodules.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80 years, regardless of gender;
* Peripheral pulmonary nodules, planned for single lesion non-anatomical sublobar resection via thoracoscopic assistance after preoperative discussion;
* Preoperative assessment indicates that the pulmonary nodules cannot be localized through visual inspection or palpation;
* Patients are able to understand the purpose of the trial, have good compliance with examinations and follow-ups, and voluntarily participate in the clinical trial by signing an informed consent form.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from this study:

- Surgical contraindications that do not meet surgical tolerance standards: fulfilling one major criterion and/or two or more minor criteria.

Major criterion: Forced expiratory volume in 1 second (FEV1) or carbon monoxide diffusion capacity (DLCO) ≤ 50%.

Minor criterion: (1) FEV1 or DLCO 51%-60%; (2) Age ≥ 75 years; (3) Pulmonary hypertension > 40 mmHg (1 mmHg = 0.133 kPa); (4) Left ventricular ejection fraction (LVEF) ≤ 40%; (5) Arterial blood partial pressure of oxygen (PaO2) < 55 mmHg or arterial blood oxygen saturation (SpO2) ≤ 88% with arterial blood partial pressure of carbon dioxide (PaCO2) > 45 mmHg.

* Contraindications for bronchoscopy, including: active massive hemoptysis; recent myocardial infarction or unstable angina; severe hypertension and arrhythmias; uncorrectable bleeding tendencies (such as severe coagulopathy, uremia, and severe pulmonary hypertension, etc.); severe superior vena cava syndrome; suspected aortic aneurysm; multiple pulmonary bullae; extremely poor overall condition;
* Female patients who are breastfeeding, pregnant, or trying to conceive;
* Patients with electromagnetic active implantable devices;
* Participants allergic to indocyanine green or anesthetics; or with a history of multiple severe allergies or hereditary allergies;
* Participation in drug clinical trials in the past 3 months, or currently participating, or participation in other medical device clinical trials within the past 30 days;
* Other conditions deemed unsuitable for participation in this clinical trial by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-10 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Success rate of staining localization | During surgical procedure
  The success rate of staining localization is defined as the number of cases with successful staining divided by the total number of cases undergoing surgery (100%). Successful staining is defined as the staining marker being clearly visible during thoracoscopy, with the staining point being less than 1 centimeter away from the nodule on the pleural projection.

SECONDARY OUTCOMES:
Re-excision rate | During surgical procedure
  The re-excision rate is defined as the number of patients requiring repeat surgery due to positive margins or inability to localize the nodule in the resected specimen, divided by the total number of patients undergoing surgery (100%).
Surgery duration | During surgical procedure
  Surgery duration is defined as the time starting from the catheter's advancement through the tracheal tube or laryngeal mask to the carina until the completion of staining localization.
Length of hospital stay | From hospital admission to discharge, assessed daily throughout the hospitalization period (expected range: 1 to 30 days)
  The length of hospital stay is defined as the time from patient admission to discharge.
Incidence of complications related to staining localization | During surgical procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: With publication
Access Criteria: Interested investigators will be required to submit a formal letter of intent outlining research aims, rationale, and approach. Furthermore, documentation of local IRB approval, including a description of type of review, should be submitted with the data request.